CLINICAL TRIAL: NCT06900608
Title: Targeted Acceptance and Commitment Therapy Compared to Supportive Therapy for Depressive Symptoms: a Pilot Randomized Controlled Trial
Brief Title: Targeted ACT Compared to Supportive Therapy for Depression RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WMich
Record Dates: First submitted 2025-03-10; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Acceptance and Commitment Therapy; Supportive Therapy
MeSH Terms: interventions — Acceptance and Commitment Therapy; Therapeutics; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Supportive Therapy (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — A 6-session ACT intervention was implemented targeting Cognitive Defusion (CD) and Values-Based Activity Scheduling (VBAS). During the first 3 sessions, the therapist taught participants how to defuse from negative self-thoughts using didactic and experiential techniques and emphasized the relationship between negative thoughts and the self and learning to observe negative thoughts for what they are - thoughts, words, ideas, and evaluations. During sessions 4-6, the therapist used similar techniques to focus on behaving in meaningful ways without letting negative thoughts dictate behavior. During these VBAS sessions, the participant identified their values and worked with the therapist to decide on goals that were values-consistent, and focused on those foals without letting negative thoughts and emotions get in the way of living toward them.
  Arms: Acceptance and Commitment Therapy
Behavioral: Treatment as usual — The 6-session supportive therapy (ST) condition emphasized the exploration of feelings; helping the client to become aware of and talk about emotional experiences with no attempt to change thoughts, behaviors, or the client's experiences directly (Greenberg et al., 1998). Psychoeducation emphasized the untoward effects of not acknowledging or exploring feelings and benefits of identification and talking about feelings. The therapist used open-ended questions, reflective listening, empathy, and clarification questions. Therapists did not give advice, offer solutions, make interpretations, or disagree with/confront the client. For homework, the participants were asked to complete "awareness homework," involving monitoring of presence, intensity, and duration of emotions with no prescription to change them or do anything differently.
  Other Names: Supportive Therapy
  Arms: Supportive Therapy

SUMMARY:
Acceptance and Commitment Therapy (ACT) has demonstrated efficacy in reducing depressive symptoms, primarily compared to no treatment or minimal treatment controls. This study compared the efficacy of ACT targeting cognitive defusion (CD, 3 sessions) and values-based activity scheduling (VBAS, 3 sessions) to supportive therapy (ST). Both treatments offered six sessions, a rationale for the approach, related techniques, and homework assignments. A parallel group randomized controlled efficacy trial design was used. Participants were stratified by gender identification and depression severity and then randomly allocated, according to a predetermined sequence, 2:1 to ACT or ST. Dependent measures were collected during acute treatment (pre, mid, and post-treatment) and follow-up at one-month.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scored one SD below the mean on the RSES and BSI
* Proficiency in English
* If taking medication for psychiatric reasons, stable medication use for at least eight weeks prior to enrollment and agreement to no changes in dosing during study participation.

Exclusion Criteria:

* Receiving other forms of psychological treatment
* Meeting PDSQ Interview criteria for psychosis, panic disorder, substance use, or endorsement of significant suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2011-12-30 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Demographic Questionnaire | Pre-treatment
Rosenberg Self-Esteem Scale | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Rosenberg Self-Esteem Scale (RSES) is a 10-item scale asking participants to rate their level of agreement (on a scale 0-4) with statements describing general feelings about themselves. Higher scores represent a more positive self-evaluation. Scores range from 0 to 40.
Brief Symptom Inventory-Global Severity Index | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Brief Symptom Inventory-Global Severity Index (BSI) is a 53-item questionnaire that provides an overview of psychological symptoms and their severity. Items are endorsed on a Likert scale (0-not at all to 4-extremely) with higher scores indicating higher rates of general distress. Scores can range from 0 to 212.
Psychiatric Diagnostic Screening Questionnaire (PDSQ) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Psychiatric Diagnostic Screening Questionnaire (PDSQ) consists of a) 125 item "yes/no" screener used to assess for symptoms of 13 psychopathologies and b) semi-structured interview(s) as indicated by endorsement of scores above the cut-off on any given psychopathology subscale based on the 125-item screener. Participants whose interview for major depressive disorder was positive for 2-4 symptoms were considered to meet criteria for minor depression, while those with 5-9 symptoms were considered to meet criteria for major depressive disorder. Each "yes" indicates one symptom, with a range of 0-9 symptoms within the depressive disorder category.
Beck Depression Inventory - II (BDI) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Beck Depression Inventory - II (BDI) is a 21-item self-report scale assessing the severity of depressive symptoms. Higher scores indicate higher rates of depressive symptoms and intensity, with scores ranging from 0-63.
Acceptance and Action Questionnaire - II (AAQ-II) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Acceptance and Action Questionnaire - II (AAQ-II) is a 7-item scale measuring experiential avoidance and psychological flexibility. Each item is scored on a 1 (never true) - 7 (always true) scale with higher scores indicate greater inflexibility. Scores range from 7-49.
Automatic Thoughts Questionnaire (ATQ) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Automatic Thoughts Questionnaire (ATQ) contains 30-items measuring the frequency and believability of negative self-statements, with higher scores indicating higher frequency or believability of thoughts. Each item is scored on a 1-5 scale (ranging from "not at all" to "all the time"), with total score ranging from 30-150.
Environmental Reward Observation Scale (EROS) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Environmental Reward Observation Scale (EROS) consists of 10 items using a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree) assessing whether affect and behavior increases as a result of contact with positively rewarding activities. Higher scores indicate larger increases when in contact with positively rewarding activities. Total scores range from 10-40.
Valued Living Questionnaire (VLQ) | Pre-treatment, 3 weeks, 6 weeks/post-treatment, and 1 month after post-treatment
  The Valued Living Questionnaire (VLQ) is a 20-item self-report measure. Participants' rate, on a scale of 1-10, first the importance of values in 10 domains (e.g., family, work, education, relationships) and then the consistency of action taken towards those values during the last week. When used as an omnibus measure the VLQ is scored by taking the mean of the products of the Importance and Consistency ratings. Higher scores indicate higher consistency or higher importance of each value. Total scores can range from 10-100.